CLINICAL TRIAL: NCT01894256
Title: An Open-label, Non-randomised, Multicentre, Comparative, Phase I Study of the Pharmacokinetics, Safety and Tolerability of Olaparib Following a Single Oral 300 mg Dose to Patients With Advanced Solid Tumours and Normal Renal Function or Renal Impairment
Brief Title: Study to Assess the Blood Levels and Safety of Olaparib in Patients With Advanced Solid Tumours and Normal or Impaired Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: D0816C00006; 2013-002225-30 (EudraCT Number)
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Solid Tumours
Keywords: oncology,; cancer,; neoplasm,; anticancer drug,; pharmacokinetics,; area under curve,; olaparib,; solid tumour,; mild renal impairment,; moderate renal impairment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal renal function (Other): Patients with calculated serum creatinine clearance ≥81 mL/min (using Cockcroft-Gault equation).
  Interventions: Drug: Olaparib tablet dosing
- Mild renal impairment (Other): Patients with calculated serum creatinine clearance 51-80 mL/min (using Cockcroft-Gault equation).
  Interventions: Drug: Olaparib tablet dosing
- Moderate renal impairment (Other): Patients with calculated serum creatinine clearance 31-50 mL/min (using Cockcroft-Gault equation).
  Interventions: Drug: Olaparib tablet dosing

INTERVENTIONS:
Drug: Olaparib tablet dosing — Part A - single 300mg oral dose olaparib (administered as 2x150mg tablets) Part B - 300mg oral dose olaparib (administered as 2x150mg tablets) bd

SUMMARY:
This is a 2-part study in patients with advanced solid tumours. Part A will investigate the PK of olaparib in patients with mild or moderate renal impairment compared to patients with normal renal function; Part B will allow eligible study patients continued access to olaparib after the PK phase and will provide additional safety data.

ELIGIBILITY:
Inclusion criteria:-

For inclusion in the study as a patient with renal impairment, the following criterion must be met:

1. Patients must have stable renal impairment (moderate or mild), depending on creatinine clearance estimated using the Cockcroft-Gault equation (moderate 31 to 50 mL/min; mild 51 to 80 mL/min), for at least 2 months prior to the start of the study. For inclusion in the study as a patient with normal renal function, the following criterion must be met:
2. Calculated serum creatinine clearance greater than or equal to 81 mL/min (using Cockcroft-Gault equation). All patients must fulfil the following criteria:
3. Provision of written informed consent prior to any study specific procedures .
4. Patients must be greater than or equal to 18 and less than or equal to 75 years of age.
5. Histologically or, where appropriate, cytologically confirmed malignant solid tumour refractory or resistant to standard therapy or for which no suitable effective standard therapy exists.
6. BMI between 18-30 kg/m2.
7. Normal liver and bone marrow function measured within 28 days prior to administration of IP as defined below: Haemoglobin (Hb) greater than or equal to 10.0 g/dL, with no blood transfusions in the previous 28 days.

   Absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L. White blood cells (WBC) greater than 3 x 109/L. Platelet count greater than or equal to 100 x 109/L. Total bilirubin less than or equal to 1.5 x institutional upper limit of normal (ULN) (except in the case of Gilbert's disease).

   Aspartate aminotransferase or serum glutamic oxaloacetic transaminase (AST), alanine aminotransferase or serum glutamic pyruvic transaminase (ALT) less than or equal to 2.5 x institutional ULN unless liver metastases are present in which case it must be less than or equal to 5x ULN.
8. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
9. Patients must have a life expectancy greater than or equal to 12 weeks.
10. Evidence of non childbearing status for women of childbearing potential, or postmenopausal status: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on Day 1 of the first treatment period in Part A. Postmenopausal is defined as:

    Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments.

    Luteinising hormone and follicle-stimulating hormone levels in the postmenopausal range for women under 50 years of age.

    Radiation-induced oophorectomy with last menses greater than 1 year ago. Chemotherapy-induced menopause with greater than 1 year interval since last menses Surgical sterilisation (bilateral oophorectomy or hysterectomy).
11. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
12. Patients must be on a stable concomitant medication regimen (with the exception of electrolyte supplements), defined as no changes in medication or in dose within 2 weeks prior to start of olaparib dosing, except for bisphosphonates, denosumab and corticosteroids, which should be stable for at least 4 weeks prior to start of olaparib dosing.

Exclusion criteria:-

Patients must not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff, its agents and/or staff at the study site).
2. Previous enrolment in the present study.
3. Participation in another clinical study with an investigational medicinal product (IP) during the last 14 days (or a longer period depending on the defined characteristics of the agent used).
4. Renal transplant and end stage renal disease (ESRD) patients.
5. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 2 weeks prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases before and during the study as long as these were started at least 4 weeks prior to treatment.
6. Patients who have received or are receiving inhibitors or inducers of CYP3A4 within the washout period.
7. For Part A only, drugs which affect creatinine clearance such as cephalosporin antibiotics, ascorbic acid, trimethoprim, cimetidine and quinine should not be used within the 7 days prior to dosing with olaparib.
8. Treatment in the previous 3 months with any drug known to have a well-defined potential for hepatotoxicity (eg, halothane).
9. Persistent toxicities (greater than or equal to CTCAE Grade 2) caused by previous cancer therapy, excluding alopecia.
10. Patients with myelodysplastic syndrome/acute myeloid leukaemia.
11. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Patients with asymptomatic brain metastases or with symptomatic but stable brain metastases can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
12. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of major surgery.
13. Patients considered a poor medical risk due to a serious uncontrolled medical disorder, non malignant systemic disease, uncontrolled seizures, or active uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive bilateral interstitial lung disease on high resolution computer tomography (HRCT) scan, or any psychiatric disorder that prohibits obtaining informed consent.
14. Patients with a history of heart failure or left ventricular dysfunction.
15. Patients who have gastric, gastro-oesophageal or oesophageal cancer.
16. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders or significant gastrointestinal resection likely to interfere with the absorption of olaparib.
17. Breastfeeding women.
18. Immunocompromised patients eg, patients who are known to be serologically positive for human immunodeficiency virus (HIV).
19. Patients with known active hepatic disease (eg, hepatitis B or C).
20. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
21. Resting ECG at screening with measurable QTc greater than 470 msec at 2 or more time points within a 24 hour period or family history of long QT syndrome.
22. Clinical judgment by the investigator that the patient should not participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anitra Fielding, Study Director — AstraZeneca Senior Research Physician; Christian Rolfo, Principal Investigator — UZ Antwerpen
Locations (13):
- Belgium (5):
  - Research Site, Brussels (Jette)
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Wilrijk
- Denmark (2):
  - Research Site, Herlev
  - Research Site, København Ø
- France (2):
  - Research Site, Bordeaux
  - Research Site, Dijon
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- United Kingdom (2):
  - Research Site, Newcastle upon Tyne
  - Research Site, Surrey

REFERENCES:
- [Derived] Rolfo C, de Vos-Geelen J, Isambert N, Molife LR, Schellens JHM, De Greve J, Dirix L, Grundtvig-Sorensen P, Jerusalem G, Leunen K, Mau-Sorensen M, Plummer R, Learoyd M, Bannister W, Fielding A, Ravaud A. Pharmacokinetics and Safety of Olaparib in Patients with Advanced Solid Tumours and Renal Impairment. Clin Pharmacokinet. 2019 Sep;58(9):1165-1174. doi: 10.1007/s40262-019-00754-4. PMID 30877569

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 20 Nov 2013; last completed Part A: 27 Mar 2015. Patients were enrolled at 13 sites in 5 countries. Part A assessed PK of olaparib in patients with mild/moderate renal impairment vs normal renal function; Part B provided additional safety data. Data are presented for Part A and Part B.
Pre-assignment Details: 56 patients were enrolled into the study, of which 12 did not fulfill the eligibility criteria. Consequently, 44 patients were assigned to treatment and received at least one dose of olaparib in Part A. Forty-three of these 44 patients were assigned treatment and received at least one dose of olaparib in Part B.
Groups:
- Normal Renal Function: Patients with calculated serum creatinine clearance ≥81 mL/min (using Cockcroft-Gault equation). Received single dose of 300 mg olaparib (2 x 150 mg tablets) in fasted condition (1 hour before their olaparib dose until 2 hours after dosing).
- Mild Renal Impairment: Patients with stable renal impairment with calculated serum creatinine clearance 51 to 80 mL/min (using Cockcroft-Gault equation), for at least 2 months prior to the start of the study.
  Received single dose of 300 mg olaparib (2 x 150 mg tablets) in fasted condition (1 hour before their olaparib dose until 2 hours after dosing).
- Moderate Renal Impairment: Patients with stable renal impairment with calculated serum creatinine clearance 31 to 50 mL/min (using Cockcroft-Gault equation), for at least 2 months prior to the start of the study.
  Received single dose of 300 mg olaparib (2 x 150 mg tablets) in fasted condition (1 hour before their olaparib dose until 2 hours after dosing).
Period: Part A
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Started | 15 | 15 | 14
Completed | 15 | 14 | 14
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Part B
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Started | 15 | 14 | 14
Completed | 0 | 0 | 0
Not Completed | 15 | 14 | 14
Not completed — Death | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lack of Efficacy | 15 | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Total
Number analyzed (Participants) | 15 | 15 | 14 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (9.90) | 63.5 (6.92) | 65.4 (12.86) | 61.9 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 7 | 25
  Male | 5 | 7 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 14 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 15 | 14 | 14 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Olaparib
Description: Maximum plasma drug concentration of olaparib
Time Frame: Part A: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK analysis set: All patients who receive an olaparib dose and have full PK sampling up to 96 hours post-dose.
  Any patients with major protocol deviations that affected the evaluability of the PK profile were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 12 | 13 | 13
μg/mL | 7.227 (31.0) | 9.081 (40.6) | 9.977 (44.2)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Null hypothesis: There are no clinically significant differences in the PK of olaparib when administered to patients with moderate or mild renal impairment compared to patients with normal renal function; Test type: Superiority or Other; Geometric least squares means ratio = 1.15, 90% CI 2-sided [1.04 to 1.27] — GLS mean for Mild Renal Impairment group vs GLS mean for Normal Renal Function
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric least squares means ratio = 1.26, 90% CI 2-sided [1.06 to 1.48] — GLS mean for Moderate Renal Impairment group vs GLS mean for Normal Renal Function

2. Primary Outcome: AUC of Olaparib
Description: Area under plasma concentration-time curve from zero to infinity of olaparib
Time Frame: Part A: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 12 | 13 | 13
μg*h/mL | 43.70 (50.1) | 70.56 (75.6) | 76.44 (78.2)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric least squares means ratio = 1.24, 90% CI 2-sided [1.06 to 1.47] — GLS mean for Mild Renal Impairment group vs GLS mean for Normal Renal Function
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric least squares means ratio = 1.44, 90% CI 2-sided [1.10 to 1.89] — GLS mean for Moderate Renal Impairment group vs GLS mean for Normal Renal Function

3. Primary Outcome: AUC0-t of Olaparib
Description: Area under plasma concentration-time curve from zero to the last measurable time point of olaparib
Time Frame: Part A: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 12 | 13 | 13
μg*h/mL | 39.97 (48.3) | 62.80 (70.3) | 69.19 (71.6)

4. Primary Outcome: Tmax of Olaparib
Description: Time to reach maximum plasma concentration of olaparib
Time Frame: Part A: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 12 | 13 | 13
Hours | 1.99 [1.07 to 3.03] | 1.55 [1.00 to 3.00] | 2.00 [1.00 to 3.00]

5. Primary Outcome: Vz/F of Olaparib
Description: Apparent volume of distribution of olaparib
Time Frame: Part A: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 12 | 13 | 13
L | 283.4 (177.9) | 131.2 (118.9) | 125.7 (167.2)

6. Primary Outcome: CL/F of Olaparib
Description: Apparent plasma clearance of olaparib
Time Frame: Part A: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 12 | 13 | 13
L/hour | 7.598 (3.649) | 5.285 (3.876) | 4.788 (2.904)

7. Primary Outcome: CLR of Olaparib
Description: Renal clearance of olaparib, calculated as the ratio of amount of drug excreted over 24 hours to AUC0-24
Time Frame: Part A: Day 1, 0-12 hours and 12-24 hours post-dose
Population: Subset of PK analysis set with urine samples available. PK analysis set: All patients who receive an olaparib dose and have full PK sampling up to 96 hours post-dose.
  Any patients with major protocol deviations that affected the evaluability of the PK profile were excluded.
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 7 | 8 | 7
L/hour | 1.4810 (0.4848) | 0.6137 (0.2859) | 0.2989 (0.1746)

8. Primary Outcome: t1/2 of Olaparib
Description: Terminal half-life of olaparib
Time Frame: Part A: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 12 | 13 | 13
Hours | 24.26 (9.749) | 17.45 (8.035) | 16.09 (9.384)

9. Other Pre Specified Outcome: Protein Binding of Olaparib
Description: Degree to which olaparib binds to the proteins within blood plasma
Time Frame: Part A: Day 1, 1 hour post-dose
Population: Subset of PK analysis set with protein binding blood sample available. PK analysis set: All patients who receive an olaparib dose and have full PK sampling up to 96 hours post-dose.
  Any patients with major protocol deviations that affected the evaluability of the PK profile were excluded.
Measure: Mean (Standard Deviation); unit: % plasma
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 13 | 12 | 14
% plasma | 7.593 (3.447) | 6.530 (2.102) | 8.022 (3.996)

10. Other Pre Specified Outcome: Free Cmax of Olaparib
Description: Cmax of unbound olaparib; calculated by multiplying total Cmax value by estimated protein binding
Time Frame: Part A: Day 1, 1 hour post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 11 | 11 | 13
μg/mL | 0.4604 (60.0) | 0.5904 (40.4) | 0.7296 (37.1)

11. Other Pre Specified Outcome: Free AUC of Olaparib
Description: AUC of unbound olaparib; calculated by multiplying total AUC by estimated protein binding
Time Frame: Part A: Day 1, 1 hour post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 11 | 11 | 13
μg*h/mL | 2.819 (65.6) | 4.771 (58.5) | 5.590 (52.2)

12. Other Pre Specified Outcome: CL/F of Unbound Olaparib
Description: Calculated from dose divided by free AUC
Time Frame: Part A: Day 1, 1 hour post-dose
Population: as for outcome 9
Measure: Median (Standard Deviation); unit: L/hour
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment
Number analyzed (Participants) | 11 | 11 | 13
L/hour | 127.7 (92.09) | 71.41 (37.40) | 59.95 (29.73)

ADVERSE EVENTS:
Time Frame: AEs were reported with an onset date between the date of first dose in the appropriate Part and the day before first dose in Part B (for Part A), or 30 days following the date of last dose of study medication if the subject discontinued (for Part B).
Description: AE data were collected on Days 1-5, and at 30 days following the date of last dose of study medication if the subject discontinued in Part A.
Groups:
- Part A Normal Renal Function: Patients from Part A of the study with calculated serum creatinine clearance ≥81 mL/min (using Cockcroft-Gault equation). Received single dose of 300 mg olaparib (2 x 150 mg tablets) in fasted condition (1 hour before their olaparib dose until 2 hours after dosing).
- Part A Mild Renal Impairment: Patients in Part A of the study with stable renal impairment with calculated serum creatinine clearance 51 to 80 mL/min (using Cockcroft-Gault equation), for at least 2 months prior to the start of the study.
  Received single dose of 300 mg olaparib (2 x 150 mg tablets) in fasted condition (1 hour before their olaparib dose until 2 hours after dosing).
- Part A Moderate Renal Impairment: Patients in Part A of the study with stable renal impairment with calculated serum creatinine clearance 31 to 50 mL/min (using Cockcroft-Gault equation), for at least 2 months prior to the start of the study.
  Received single dose of 300 mg olaparib (2 x 150 mg tablets) in fasted condition (1 hour before their olaparib dose until 2 hours after dosing).
- Part B Normal Renal Function: Patients in Part B of the study with calculated serum creatinine clearance ≥81 mL/min (using Cockcroft-Gault equation). Received single dose of 300 mg olaparib (2 x 150 mg tablets) in fasted condition (1 hour before their olaparib dose until 2 hours after dosing).
- Part B Mild Renal Impairment: Patient in Part B of the study with stable renal impairment with calculated serum creatinine clearance 51 to 80 mL/min (using Cockcroft-Gault equation), for at least 2 months prior to the start of the study.
  Received single dose of 300 mg olaparib (2 x 150 mg tablets) in fasted condition (1 hour before their olaparib dose until 2 hours after dosing).
- Part B Moderate Renal Impairment: Patient in Part B of the study with stable renal impairment with calculated serum creatinine clearance 31 to 50 mL/min (using Cockcroft-Gault equation), for at least 2 months prior to the start of the study.
  Received single dose of 300 mg olaparib (2 x 150 mg tablets) in fasted condition (1 hour before their olaparib dose until 2 hours after dosing).
Arm/Group | Part A Normal Renal Function | Part A Mild Renal Impairment | Part A Moderate Renal Impairment | Part B Normal Renal Function | Part B Mild Renal Impairment | Part B Moderate Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 0/14 | 3/15 | 3/14 | 3/14
Other Adverse Events (participants affected / at risk) | 10/15 | 11/15 | 6/14 | 15/15 | 14/14 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Normal Renal Function (N=15) | Part A Mild Renal Impairment (N=15) | Part A Moderate Renal Impairment (N=14) | Part B Normal Renal Function (N=15) | Part B Mild Renal Impairment (N=14) | Part B Moderate Renal Impairment (N=14)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
ILEUS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
NON CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
UROSEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Normal Renal Function (N=15) | Part A Mild Renal Impairment (N=15) | Part A Moderate Renal Impairment (N=14) | Part B Normal Renal Function (N=15) | Part B Mild Renal Impairment (N=14) | Part B Moderate Renal Impairment (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 2 | 3 | 5 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 2 | 2
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 4 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 2 | 0 | 9 | 7 | 8
VOMITING (Gastrointestinal disorders) | 1 | 2 | 0 | 4 | 5 | 4
ASTHENIA (General disorders) | 0 | 1 | 1 | 2 | 2 | 3
FATIGUE (General disorders) | 1 | 0 | 1 | 8 | 8 | 8
PYREXIA (General disorders) | 1 | 1 | 0 | 1 | 4 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 3
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
ALTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 1 | 0 | 1 | 3 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 2
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 4 | 2 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 5 | 1 | 3
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 6 | 4
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 2
NON CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 1 | 2 | 2
ODEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 2 | 4 | 1
WEIGHT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 3
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 5 | 5
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 1 | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 3 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 3 | 2 | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Data are presented for Part A and Part B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other